CLINICAL TRIAL: NCT04363281
Title: The Effect of Anxiety on Perioperative Pain: Patient and Provider Perception : A Prospective Observational Study
Brief Title: The Effect of Anxiety on Perioperative Pain: Patient and Provider Perception
Status: Completed | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, sharonorbach, Professor Sharon Orbach-Zinger, Rabin Medical Center
Other Study IDs: 409-19
Record Dates: First submitted 2020-02-13; First posted 2020-04-27 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: preoperative questionnaire — 1. Three questions to predict acute pain:
     * Verbal numeric score Anxiety 0-10
     * Anticipated postoperative pain level
     * Anticipated analgesic requirements
  2. Speilberger STATE-TRATE inventory index
  3. Pain Catastrophizing Scale
Other: PACU questionnaire — parturients will be approached and requested to fill out a questionnaire regarding intraoperative pain, medication consumption, anxiety and nausea.
Other: Postoperative questionnaire — Parturients will be approached at 24 hours postpartum and questioned regarding anxiety levels and medication consumption and requested to fill out the OBSQOR 11 questionnaire at 24 hours postpartum.
Other: Postoperative questionnaire- Obstetrician — The attended obstetrician will be questioned regarding the parturient's level of intraoperative pain, postoperative pain levels anxiety medication consumption, uteronic management, surgical technique and management.
Other: Postoperative questionnaire- anesthesiologist — he attended anesthesiologist will be questioned regarding the parturient's level of intraoperative pain, postoperative pain levels anxiety medication consumption, uteronic management, surgical technique and management.

SUMMARY:
In this study we will assess the incidence and severity of intraoperative and postoperative pain and determine the effect of preoperative anxiety on intraoperative and postoperative pain incidence. Secondary outcome is to assess provider perception of pain.

DETAILED DESCRIPTION:
This is a prospective, observational study. Following obtaining written formal consent parturients will be requested to fill out the following questionnaires

1. Three questions to predict acute pain:

   * Verbal numeric score Anxiety 0-10
   * Anticipated postoperative pain level
   * Anticipated analgesic requirements
2. Speilberger STATE-TRATE inventory index
3. Pain Catastrophizing Scale In the post anesthesia care unit (PACU) parturients will be approached and requested to fill out a questionnaire regarding intraoperative pain, medication consumption, anxiety and nausea. Furthermore parturients will also be approached at 12 hours and 48 hours postpartum and questioned regarding anxiety levels and medication consumption and requested to fill out the OBSQOR 11 questionnaire at 12 hours postpartum.

Additionally, both the attending anesthesiologist and obstetrician will be questioned regarding the parturient's level of intraoperative pain, postoperative pain levels anxiety medication consumption, uteronic management, surgical technique and management.

ELIGIBILITY:
Inclusion Criteria:

*Women undergoing an elective cesarean section under spinal anesthesia with the ability to comply with the study requirements will be eligible for participation

Exclusion Criteria:

* All women unable to receive spinal anesthesia or with inadequate spinal anesthesia prior to the beginning of surgery (Less than T4 Sensory Level to pinprick assessed from blunt tip needle in caudal to cranial direction )
* All women receiving antianxiety medication
* Language barrier

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Parturients will be approached and consented for participation in the women's surgery unit on the day of surgery when they aren't under any pain or sedatives.
Sampling Method: Non-Probability Sample
Enrollment: 193 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Verbal numeric Score of postoperative pain | 24 hours
  measured by a verbal numeric score from 0-10
Verbal numeric Score of intraoperative pain | 1 hour during surgery
  measured by a verbal numeric score from 0-10
Preoperative Anxiety | 2 hours before surgery
  Score from 0-10

SECONDARY OUTCOMES:
Patient provider perception of pain | 1 hour during surgey
  measured by a verbal numeric score from 0-10

CONTACTS AND LOCATIONS:
Locations (1):
- Beilinson hospital, Petach Tikvah, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bierke S, Petersen W. Influence of anxiety and pain catastrophizing on the course of pain within the first year after uncomplicated total knee replacement: a prospective study. Arch Orthop Trauma Surg. 2017 Dec;137(12):1735-1742. doi: 10.1007/s00402-017-2797-5. Epub 2017 Sep 30. PMID 28965133
- [Background] Raichle KA, Osborne TL, Jensen MP, Ehde DM, Smith DG, Robinson LR. Preoperative state anxiety, acute postoperative pain, and analgesic use in persons undergoing lower limb amputation. Clin J Pain. 2015 Aug;31(8):699-706. doi: 10.1097/AJP.0000000000000150. PMID 26153780
- [Background] Aouad MT, Kanazi GE, Malek K, Tamim H, Zahreddine L, Kaddoum RN. Predictors of postoperative pain and analgesic requirements following abdominal hysterectomy: an observational study. J Anesth. 2016 Feb;30(1):72-9. doi: 10.1007/s00540-015-2090-0. Epub 2015 Oct 24. PMID 26499321
- [Background] Ip HY, Abrishami A, Peng PW, Wong J, Chung F. Predictors of postoperative pain and analgesic consumption: a qualitative systematic review. Anesthesiology. 2009 Sep;111(3):657-77. doi: 10.1097/ALN.0b013e3181aae87a. PMID 19672167
- [Background] Gorkem U, Togrul C, Sahiner Y, Yazla E, Gungor T. Preoperative anxiety may increase postcesarean delivery pain and analgesic consumption. Minerva Anestesiol. 2016 Sep;82(9):974-80. Epub 2016 Mar 30. PMID 27028449
- [Background] Pan PH, Tonidandel AM, Aschenbrenner CA, Houle TT, Harris LC, Eisenach JC. Predicting acute pain after cesarean delivery using three simple questions. Anesthesiology. 2013 May;118(5):1170-9. doi: 10.1097/ALN.0b013e31828e156f. PMID 23485992
- [Background] McCombe K, Bogod DG. Learning from the Law. A review of 21 years of litigation for pain during caesarean section. Anaesthesia. 2018 Feb;73(2):223-230. doi: 10.1111/anae.14119. Epub 2017 Nov 1. PMID 29090735